CLINICAL TRIAL: NCT04870905
Title: Tisleilizumab (PD-1 Antibody) and Chemoradiotherapy in Locoregionally-advanced Nasopharyngeal Carcinoma: a Phase 2 Trial
Brief Title: Tisleilizumab (PD-1 Antibody) and Chemoradiotherapy in Locoregionally-advanced Nasopharyngeal Carcinoma
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Affiliated Cancer Hospital & Institute of Guangzhou Medical University (Other)
Collaborators: Union hospital of Fujian Medical University (Other); Zhujiang Hospital (Other); Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, Yuan yawei, Professor, Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICRT-001
Record Dates: First submitted 2021-05-01; First posted 2021-05-04 (Actual); Last update posted 2023-03-06 (Actual); Status verified 2023-03

CONDITIONS: Nasopharyngeal Neoplasms
MeSH Terms: conditions — Nasopharyngeal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICRT arm (Experimental)
  Interventions: Drug: Tis-U-Sol

INTERVENTIONS:
Drug: Tis-U-Sol — Tislelizumab 200mg will be given every 3 weeks for 12 cycles

SUMMARY:
This trial intends to enroll patients with T4N1 or T1-4N2-3 (AJCC 8th) locoregionally-advanced nasopharyngeal carcinoma (LANPC). All the Patients will receive 3 cycles of induction chemotherapy with docetaxel and cisplatin and cisplatin based concurrent chemoradiotherapy (CCRT) plus adjuvant immunotherapy (tisleilizumab). All patients will receive intensity-modulated radiotherapy (IMRT). Tisleilizumab will begin 4-6 weeks after CCRT and continue every 3 weeks for 12 cycles.

ELIGIBILITY:
Inclusion Criteria:

- Patients with histologically confirmed nasopharyngeal carcinoma. Stage T4N1 or T1-4N2-3 (AJCC 8th). Eastern Cooperative Oncology Group performance status ≤1. Adequate marrow function: neutrocyte count≥1.5×10e9/L, hemoglobin ≥90g/L and platelet count ≥100×10e9/L.

Alanine Aminotransferase (ALT)/Aspartate Aminotransferase (AST) ≤2.5×upper limit of normal (ULN), and bilirubin ≤ 1.5×ULN.

Adequate renal function: creatinine clearance rate ≥ 60 ml/min (Cockcroft-Gault formula).

Patients must be informed of the investigational nature of this study and give written informed consent.

Women of childbearing potential (WOCBP) who are sexually active must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of study drug. Men who are sexually active with WOCBP must be willing to adhere to effective contraception during treatment and for 1 year after the last dose of the study drug.

Exclusion Criteria:

Hepatitis B surface antigen (HBsAg) positive and hepatitis B virus DNA >1×10e3 copies/ml or 200IU/ml;Hepatitis C virus (HCV) antibody positive Has active autoimmune disease, except type I diabetes, hypothyroidism treated with replacement therapy, and skin disease that doesn't require systemic treatment (e.g., vitiligo, psoriasis, or alopecia).

Has any condition that required systemic corticosteroid (equivalent to prednisone >10mg/d) or other immunosuppressive therapy within 28 days before informed consent. Patients received systemic corticosteroid equivalent to prednisone ≤10mg/d, inhale or topical corticosteroid will be allowed.

Has a known history of active TB (bacillus tuberculosis) within 1 year; patients with adequately treated active TB over 1 year ago will be allowed.

Has a known history of interstitial lung disease. Heart disease that is not well controlled,including symptomatic heart failure, unstable angina, myocardial infarction.

Is pregnant or breastfeeding. Prior malignancy within 5 years, except in situ cancer, adequately treated non-melanoma skin cancer, and papillary thyroid carcinoma.

Has known allergy to large molecule protein products or any compound of tisleilizumab.

Has a known history of human immunodeficiency virus (HIV) infection. Active infection requiring systemic therapy. A history of psychotropic substance abuse, alcohol or drug abuse Any other condition, including mental illness or domestic/social factors, deemed by the investigator to be likely to interfere with a patient's ability to sign informed consent, cooperate and participate in the study, or interferes with the interpretation of the results.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Failure-free survival (FFS) | 3 years
  From randomization to the date of locoregional failure, distant failure, or death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Principal investigator Principal investigator, Principal Investigator — Affiliated Cancer Hospital & Institute of Guangzhou Medical University
Locations (1):
- Affiliated Cancer Hospital & Institute of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lee AW, Ngan RK, Tung SY, Cheng A, Kwong DL, Lu TX, Chan AT, Chan LL, Yiu H, Ng WT, Wong F, Yuen KT, Yau S, Cheung FY, Chan OS, Choi H, Chappell R. Preliminary results of trial NPC-0501 evaluating the therapeutic gain by changing from concurrent-adjuvant to induction-concurrent chemoradiotherapy, changing from fluorouracil to capecitabine, and changing from conventional to accelerated radiotherapy fractionation in patients with locoregionally advanced nasopharyngeal carcinoma. Cancer. 2015 Apr 15;121(8):1328-38. doi: 10.1002/cncr.29208. Epub 2014 Dec 19. PMID 25529384
- [Background] Lv X, Cao X, Xia WX, Liu KY, Qiang MY, Guo L, Qian CN, Cao KJ, Mo HY, Li XM, Li ZH, Han F, He YX, Liu YM, Wu SX, Bai YR, Ke LR, Qiu WZ, Liang H, Liu GY, Miao JJ, Li WZ, Lv SH, Chen X, Zhao C, Xiang YQ, Guo X. Induction chemotherapy with lobaplatin and fluorouracil versus cisplatin and fluorouracil followed by chemoradiotherapy in patients with stage III-IVB nasopharyngeal carcinoma: an open-label, non-inferiority, randomised, controlled, phase 3 trial. Lancet Oncol. 2021 May;22(5):716-726. doi: 10.1016/S1470-2045(21)00075-9. Epub 2021 Apr 12. PMID 33857411
- [Background] Chen YP, Chan ATC, Le QT, Blanchard P, Sun Y, Ma J. Nasopharyngeal carcinoma. Lancet. 2019 Jul 6;394(10192):64-80. doi: 10.1016/S0140-6736(19)30956-0. Epub 2019 Jun 6. PMID 31178151
- [Background] Zhang Y, Chen L, Hu GQ, Zhang N, Zhu XD, Yang KY, Jin F, Shi M, Chen YP, Hu WH, Cheng ZB, Wang SY, Tian Y, Wang XC, Sun Y, Li JG, Li WF, Li YH, Tang LL, Mao YP, Zhou GQ, Sun R, Liu X, Guo R, Long GX, Liang SQ, Li L, Huang J, Long JH, Zang J, Liu QD, Zou L, Su QF, Zheng BM, Xiao Y, Guo Y, Han F, Mo HY, Lv JW, Du XJ, Xu C, Liu N, Li YQ, Chua MLK, Xie FY, Sun Y, Ma J. Gemcitabine and Cisplatin Induction Chemotherapy in Nasopharyngeal Carcinoma. N Engl J Med. 2019 Sep 19;381(12):1124-1135. doi: 10.1056/NEJMoa1905287. Epub 2019 May 31. PMID 31150573
- [Background] Sun Y, Li WF, Chen NY, Zhang N, Hu GQ, Xie FY, Sun Y, Chen XZ, Li JG, Zhu XD, Hu CS, Xu XY, Chen YY, Hu WH, Guo L, Mo HY, Chen L, Mao YP, Sun R, Ai P, Liang SB, Long GX, Zheng BM, Feng XL, Gong XC, Li L, Shen CY, Xu JY, Guo Y, Chen YM, Zhang F, Lin L, Tang LL, Liu MZ, Ma J. Induction chemotherapy plus concurrent chemoradiotherapy versus concurrent chemoradiotherapy alone in locoregionally advanced nasopharyngeal carcinoma: a phase 3, multicentre, randomised controlled trial. Lancet Oncol. 2016 Nov;17(11):1509-1520. doi: 10.1016/S1470-2045(16)30410-7. Epub 2016 Sep 27. PMID 27686945
- [Background] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452